CLINICAL TRIAL: NCT00352209
Title: Retrospective Review of Cardiomyopathy Patient Cases Post Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Cardiomyopathy Following Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060158; 06-CC-0158
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-05-16

CONDITIONS: Cardiomyopathy
Keywords: Cyclophosphamide; Preparative Regimens; Risk Factors; Chart Review; Incidence
MeSH Terms: conditions — Cardiomyopathies

SUMMARY:
This study will examine the incidence of cardiac complications, particularly cardiomyopathy, in patients who have undergone allogeneic (donor) stem cell transplantation at NIH. Cardiac complications in these patients are well documented. Most commonly, patients develop congestive heart failure or pericarditis after receiving high-dose cyclophosphamide, radiation, or other intensive chemotherapy regimens prior to the transplant.

Most data in the medical literature suggest that the rate of serious cardiac complications is relatively low, at about 5 percent or less. Recently, a cluster of cases of significant cardiomyopathy in stem cell transplant patients at the NIH Clinical Center has prompted concern that the incidence of these complications is higher than that reported in the medical literature.

This study will further define the incidence of cardiac problems, primarily focusing on cardiomyopathy, with the following objectives:

* To define the incidence of cardiomyopathy in allogeneic stem cell transplant patients enrolled in National Cancer Institute (NCI) and National Heart, Lung, and Blood (NHLBI) protocols at the NIH Clinical Center
* To document the presence or absence of various known or suspected risk factors for cardiomyopathy in the documented cases.

The study consists of a chart review of patients who have had an allogeneic stem cell transplant on either an NHLBI or NCI protocol since 1999.

This project is a first step in clarifying the cardiac complications following stem cell transplantation, their incidence, and characteristics of the patient populations. It will look at patient demographics, the characteristics of the cardiac complication, and known or suspected risk factors.

DETAILED DESCRIPTION:
Cardiac complications in patients who have undergone allogeneic hematopoietic stem cell transplantation (HSCT) have been well documented. Most commonly patients present with congestive heart failure and/or pericarditis after receiving high-dose cyclophosphamide, total body irradiation (TBI) or other intensive conditioning / preparative regimens prior to the allogeneic transplant. The majority of the data in the medical literature suggests that the rate of serious cardiac events appears to be relatively low at approximately 5% or less. Recently, there appears to have been a cluster of patient cases (approximately 15) of significant cardiomyopathy in patients who have received an allogeneic HSCT at the NIH Clinical Center over the past year. These cases have been consulted on by the Cardiology consult service and have included both NCI and NHLBI protocol patients. This cluster of cases has prompted concern that the incidence of cardiac toxicity recently seen at the NIH Clinical Center is not consistent with the reported incidence of significant cardiac toxicity in the medical literature.

The proposed retrospective chart review is intended to further define the incidence of cardiac toxicity, primarily focusing on cardiomyopathy. The project is an initial step to consolidate the data from both the NCI and NHLBI transplant programs and clarify the documented cardiac toxicities, the incidence, and the demographics of the patient populations. We also plan to document the presence or absence of a variety of known and suspected risk factors for cardiotoxicity. This analysis will only be preliminary but will potentially lead to more formal prospective studies on cardiotoxicity related to allogeneic HSCT.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Patients who have undergone an allogeneic HSCT on either an NHLBI or NCI protocol since 1999 will be the patient population for this chart review. Patients with documented serious cardiac events will be identified from NHLBI cardiology consult records, NCI and NHLBI research data bases, and the data base of the echocardiogram service.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-05-02; Study Completion 2007-05-16

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Heart, Lung and Blood Institute (NHLBI), 9000 Rockville Pike, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Goldberg MA, Antin JH, Guinan EC, Rappeport JM. Cyclophosphamide cardiotoxicity: an analysis of dosing as a risk factor. Blood. 1986 Nov;68(5):1114-8. PMID 3533179